CLINICAL TRIAL: NCT01594151
Title: Modelling of the Upper Airway in Children With Controlled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FLUI-2010-59; 2011-000286-12 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Controlled Asthma
Keywords: asthma; controlled; Cone Beam Computed Tomography; upper airway; paediatric
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography — CBCT scan of upper airway at visit 1
  Other Names: CBCT

SUMMARY:
Asthma in children is recognized as a disease area with a high medical need. As the investigators move into this field it is necessary to improve the investigators knowledge of upper airway anatomical structure in paediatric patients. This study will provide airway/facial morphologies from controlled asthmatic patients. Limited facial morphology can be used in order to build models to study the delivery of medication through a device that requires for example a facemask. In this study the anatomical structure of the upper airway and the facial geometry will be evaluated using a Cone Beam Computed Tomography (CBCT) scan. The scan will be taken in a population of 20 asthmatic children between 6 and 12 years old.

ELIGIBILITY:
Inclusion Criteria:

* Male and pre-menarchial female children aged 6-12yrs on visit 1. Pre-menarchial females are defined in this study as girls with breast stage 1 or 2 and no menarche.
* Parents or guardian must be able to understand and complete to protocol requirements, instructions and protocol-stated restrictions. Parents/guardians must give written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Diagnosis of asthma at least 6 months previous prior to screening.
* Children must be controlled on their existing asthma treatment at screening as defined by ACT or childhood ACT score of ≥ 20 and PEF>80%.
* Children must be taking a stable regime of SABA/ LABA on an as need basis, with or without Leukotriene Antagonists and inhalation corticosteroids.
* All children must be competent to perform the required tests.
* Children must be available to complete the study and comply with study primary objective investigations.
* Children must be able to withhold from short acting bronchodilators for 6 hours.

Exclusion Criteria:

* As a result of the medical interview, physical examination or screening investigations, the responsible physician considers the patient unsuitable for inclusion to the study.
* Children who have a past or present disease, or have had previous surgery which as judged by the Investigator, may affect patient safety or influence the outcome of the study.
* The child has received an investigational drug or participated in any other research trial within 30 days, or twice the duration of the biological effect of any drug (whichever is longer).
* The child has had a respiratory tract infection within two weeks of the start of the study.
* Children who have had an exacerbation of disease requiring hospitalization for > 24 hrs within four weeks prior to inclusion.
* Children who are unwilling or unable to follow any of the procedures outlined in the protocol.
* Child is mentally incapacitated.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cone Beam Computed Tomography | At day 1
  The primary objective of this study is to provide data from CBCT scans to evaluate the anatomical structure of the upper airway and the facial geometry of children. The provided data will enable further work in the mapping of the upper airway and deliver 3D geometries.

CONTACTS AND LOCATIONS:
Overall Officials: Désirée van Doorn, MD, Principal Investigator — Heilig Hart Hospital Lier
Locations (1):
- Private Practice Dr. van Doorn, Kontich, Antwerp, Belgium